CLINICAL TRIAL: NCT05341791
Title: Comparing Novel Methods of Study Information Notice Administration to the Standard Approach in Enhancing Clinical Studies Understanding in Resource Limited Settings: A Randomized Trial
Brief Title: Paper Versus Cartoon Video-based Administration of Study Information Notice for Participant Consent
Acronym: CONSENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EG0266
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Information Disclosure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard administration of information notice (No Intervention): : During the standard study information administration, the participant will read though the written information notice which will be organized in sections. After each section, the study staff will explain to the participant the key information to understand. Throughout the process, participants will be allowed to ask study staff questions. We anticipate the time to administer consent by this standard approach will be approximately 45 to 60 minutes per participants.
- video administration of information notice (Experimental): The video will be 20-minutes long, and will consist of graphic depictions (in cartoon style) of the study information content presented in the same flow as the written notice, and explained by a voice-over in the background. The participant will view the video in a quiet room, on a tablet provided by the study staff. The participant will be able to pause the video or rewind it as needed, and view it at his/her desired pace. The video will have an embedded knowledge check at the end of each section, consisting of a background voice asking some questions, pausing (for the participant to think through the correct answers) and then providing the right answers.
  Interventions: Other: Cartoon video describing study information notice

INTERVENTIONS:
Other: Cartoon video describing study information notice — The video will be 20-minutes long, and will consist of graphic depictions (in cartoon style) of the study information content presented in the same flow as the written notice, and explained by a voice-over in the background. The participant will view the video in a quiet room, on a tablet provided by the study staff. The participant will be able to pause the video or rewind it as needed, and view it at his/her desired pace. The video will have an embedded knowledge check at the end of each section, consisting of a background voice asking some questions, pausing (for the participant to think through the correct answers) and then providing the right answers.
  Arms: video administration of information notice

SUMMARY:
This study is a randomized trial in which participants are assigned to one of 2 strategies of information notice administration which include the standard approach versus a video-based cartoon approach. An information notice about the study will be administered to each participant individually. The study involves the integration of tuberculosis screening at all pediatric entry points, and other activities aimed at improving pediatric tuberculosis diagnosis and management. The understanding of participants will be assessed using a test of understanding adapted from the Quality of Informed consent (QIC).

DETAILED DESCRIPTION:
Objectives:

Primary Objective: is to evaluate the effectiveness of cartoon video-based study information notice administration compared to standard study information notice administration as assessed by the QIC Secondary Objectives: - Determine the factors associated with effectiveness of the cartoon video-based study information notice administration.

Endpoints:

Primary Endpoint: The proportion of participants scoring more than 80% at the test of understanding, comparing the novel and the standard strategy.

Study Population: Our population will consist of adults bringing their children for routine care in the facilities in which the study will be conducted.

Study Sites This study will be conducted in 4 sites located in the West, Littoral and Center regions of Cameroon. These sites are the District Hospital of Dschang, the district hospital of Foumban, the District hospital of Loum, and the district hospital of Soa. These sites are semi-urban sites and are selected to facilitate inclusion of participants from urban, peri-urban and rural settings. Also, these sites conduct routine systematic and active screening for pediatric tuberculosis of all children presenting for care in the facility, as well as other interventions to improve pediatric tuberculosis diagnosis and management. These tuberculosis activities, which had been implemented by EGPAF through the CaP TB program are now part of the routine sites activities and will be used to build the information notice for the purpose of this study.

Participant's eligibility and recruitment process Eligible participants will be adults (of at least 21 years of age), or emancipated minors bringing their children (of less than 15 years) for routine care in the selected facilities, and able to read and write English or French and who accept to be part of the study. Every day, routine triage registers (and/or immunization registers, depending on the organization of the health facility) will be used to identify parents bringing their children for routine care. Parents whose children have a serial number in the register which is a multiple of 3 will be screened for eligibility to the study and enrolled if eligible and after providing a written consent. A maximum of 10 participants will be enrolled per day. All enrolled participants will be randomly allocated to the intervention arm (video-cartoon) or to standard consenting following a 1:1 ratio.

Description of the information notice to be administered An information notice on the integration of tuberculosis activities at all pediatric entry points will be developed. This information notice will include details on definition of tuberculosis, rationale and process of systematic and active screening for tuberculosis at all pediatric entry points, sample collection and chest X-ray procedures and indications, data collected as part of the TB activities in the sites, risks and benefits of TB screening and diagnosis procedures, and possibility to accept or refuse TB procedures.

Description of Study arms:

There are 2 study arms. The standard administration of information notice consists of a paper-based study information notice which is provided to the participant during a one-to-one conversation with a study staff. The participant either reads the study information notice or it is read to him/her and explained section by section. The video-based study information notice administration consists of a 20 minutes' cartoon video explaining the study which will be played to the participant.

Study Duration: 20 months

Participant Duration in the study: 1 day

ELIGIBILITY:
Inclusion Criteria:

* All adults > = 21 years of age, or emancipated minors (persons between 15-17 years who are married or pregnant/have children or head of a household)
* Are able to speak, read and write English or French
* Bringing their children for routine consultation or immunization in the selected study sites
* Give their written consent to take part to the study

Exclusion Criteria:

- Participants with visual or hearing challenges which prevent them from reading written forms or viewing/listening to a video content will be excluded Selection of participants

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
The proportion of participants scoring more than 80% on the test of understanding, comparing the novel and the standard strategy. | 1 day
  The proportion of participants scoring more than 80% on the test of understanding, comparing the novel and the standard strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Boris K Tchounga, MD, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (1):
- HD SOA, Yaoundé, Centre Region, Cameroon

IPD SHARING:
Plan to Share IPD: No